CLINICAL TRIAL: NCT05330585
Title: Functional Near-infrared Spectroscopy (fNIRS) as a Measure of Listening Effort and Speech Intelligibility in Adults With Hearing Loss
Brief Title: fNIRs, Listening Effort, and Speech Intelligibility
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Sonova AG (Industry)
Collaborators: Toronto Metropolitan University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: SRF-1412
Record Dates: First submitted 2022-04-08; First posted 2022-04-15 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-03

CONDITIONS: Hearing Loss
MeSH Terms: conditions — Hearing Loss | interventions — Hearing Aids

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participants with hearing loss. (Experimental): Participants with hearing loss.
  Interventions: Device: Hearing aids; Other: Unaided

INTERVENTIONS:
Device: Hearing aids — Participants will listen to stimuli in the environment while wearing hearing aids which should make the stimuli more audible. Speech in noise performance is expected to improve and PFC oxygenation is expected to be reduced in this condition.
  Other Names: Investigational
Other: Unaided — Participants will listen to stimuli in the environment with their hearing loss. Speech in noise performance is expected to decline and PFC oxygenation is expected to be increased in this condition.
  Other Names: Control

SUMMARY:
The purpose of the current study is to measure oxygenation in the PFC using fNIRS in a sample of older adults with hearing loss. Adults with hearing loss will be asked to repeat the final word from low-context sentences in noise at two SNRs; a hard SNR (individually-measured SNR-50), and an easy SNR (SNR-50 + 10 dB) both without and with hearing aids set to a directional mode. The procedure will be a within-subject repeated measures. Stimuli will be randomized.

DETAILED DESCRIPTION:
See above.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18-99 years) with ≥3 months hearing aid experience
* binaural, symmetric, sensorineural N2 (mild) to N6 (severe) hearing loss
* fluent in English

Exclusion Criteria:

* children/teenagers
* normal hearing or hearing loss exceeding N6 (severe) by 10 dB

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-05-03 (Actual); Primary Completion 2022-11 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Listening effort | Up to 2 hours during 1 session
  Listening effort inferred from infrared light scattered from the prefrontal cortex, which is indicative of concentration of oxygenated blood in that region. A higher concentration is indicative of more listening effort.
Speech-in-noise performance | Up to 2 hours during 1 session
  Number of words repeatedly correctly for a given listening condition.

CONTACTS AND LOCATIONS:
Overall Officials: Jinyu Qian, PhD, Principal Investigator — Sonova AG
Locations (1):
- Sonova Innovation Centre Toronto, Mississauga, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No